CLINICAL TRIAL: NCT06720909
Title: Feasibility of Combining Mindfulness Intervention and Open-Label Placebo Treatment for Chronic Pain
Brief Title: Mindfulness And Placebo for Pain (MAPP) Study
Acronym: MAPP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Chung Jung Mun, Assistant Professor, Arizona State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00020051; 1R34AT012677 (NIH)
Record Dates: First submitted 2024-12-03; First posted 2024-12-06 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Chronic Pain
Keywords: chronic pain; pain; mindfulness; placebo
MeSH Terms: conditions — Chronic Pain; Pain | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- MBSR-Only (Experimental): This experimental arm receives the 8-week MBSR program only.
  Interventions: Behavioral: Mindfulness-Based Stress Reduction (MBSR)
- OLP-Only (Experimental): This experimental arm receives the OLP treatment only.
  Interventions: Other: Open-Label Placebo (OLP)
- MBSR+OLP (Experimental): This experimental arm receives the 8-week MBSR program AND the 8-week OLP treatment.
  Interventions: Other: MBSR+OLP

INTERVENTIONS:
Behavioral: Mindfulness-Based Stress Reduction (MBSR) — The standard 8-week MBSR program will be led by certified MBSR instructors from the UCSD Center for Mindfulness. The program content will consist of a variety of mindfulness and meditative techniques, such as sitting meditation, body scans, and mindful yoga. Participants will engage in weekly sessions via Zoom, participation in group discussions, and honing their other mindfulness skills. Throughout the program, participants will be instructed to commit to a daily mindfulness meditation practice lasting approximately 45 minutes, at least 6 days a week.
  Arms: MBSR-Only
Other: Open-Label Placebo (OLP) — The placebo pills will be size #1 capsules filled with (1) microcrystalline cellulose, a common inert excipient for pharmaceuticals, and (2) 25 mg riboflavin tracer. Participants will be informed that the placebo pills are inactive substances, like sugar pills, and contain no active medication. Then, they will watch a brief introduction video which will cover four main discussion points: (1) the placebo effect can be powerful and can have beneficial effects for diverse symptoms, (2) the body can respond to taking placebo pills automatically despite the knowledge that it is placebo (e.g., Pavlov's dogs), (3) a positive attitude or expectation can be beneficial but is not necessary, and (4) taking the pills faithfully throughout the intervention period is critical.
  Arms: OLP-Only
Other: MBSR+OLP — This condition involves a combination of interventions, where participants will receive both MBSR and OLP treatments.
  Arms: MBSR+OLP

SUMMARY:
This study proposes a three-arm randomized-controlled trial (RCT) that evaluates the feasibility and acceptability of combining a mindfulness-based therapy (MBT) and open-label placebo (OLP) treatment for individuals with chronic pain. Individuals with chronic pain will be recruited to participate in an 8-week trial, with a subsequent 3-month post-treatment follow-up.

Participants will be randomly assigned to one of the following three conditions:

1. Mindfulness-Based Stress Reduction (MBSR)
2. OLP treatment
3. combination of MBSR and OLP treatment

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years old;
2. ability to speak, write, and read in English;
3. physical pain present on at least half the days in the past 3 months; and
4. average past week pain severity rating ≥3 on a 0-10 Numerical Rating Scale.

Exclusion Criteria:

1. acute pain due to recent injury or surgery;
2. self-reporting of chronic malignant pain (e.g., cancer, HIV);
3. self-reporting of Raynaud's disease (those who can be contraindicated for cold pressor testing);
4. severe psychopathology (e.g., a psychotic disorder) or significant cognitive deficits judged to interfere with study procedures;
5. currently pregnant or breastfeeding;
6. inability to discontinue use of vitamin B2 supplements or a multivitamin containing vitamin B2 throughout the study period (these interfere with riboflavin tracer-OLP treatment adherence-monitoring);
7. inability to commit to study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-01-27 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Feasibility - Feasibility of Participant Enrollment | Enrollment
  Feasibility of participant enrollment will be benchmarked at 100% (N=45) proposed participant enrollment during the study.
Feasibility - Participant Retention | Enrollment to end of 3-month follow-up
  Participant retention will be benchmarked at a ≥75% retention rate from baseline to 3-month follow-up.
Feasibility - MBSR Intervention Adherence | Enrollment to end of 8-week treatment
  Intervention adherence for MBSR will be benchmarked as an average of ≥75% (6 out of 8) MBSR session completion AND and average of ≥75% daily mindfulness homework completion.
Feasibility - OLP Treatment Adherence | Enrollment to end of 8-week treatment
  Intervention adherence for OLP treatment will be benchmarked as an average of ≥75% adherence to OLP treatment based upon percent days OLP consumed measured by MEMS (Medication Event Monitoring System) SmartCap AND detection of riboflavin tracer in urine samples during both the mid- and post-treatment sessions.
Feasibility - Daily Diary Assessment Compliance | Enrollment to end of 3-month follow-up
  Daily diary assessment compliance will be benhcmarked as an average of ≥75% compliance throughout the study period including baseline, mid-treatment, post-treatment, and 3-month follow-up.
Acceptability - Global Satisfaction | Enrollment to end of 8-week treatment
  Global satisfaction will be benchmarked as an average score of ≥75 from a 0-100 scale.
Acceptability - Perceived Intervention Effectiveness | Enrollment to end of 8-week treatment
  Perceived intervention effectiveness will be benchmarked as an average score of ≥75 from a 0-100 scale.
Acceptability - Perceived Intervention Convenience | Enrollment to end of 8-week treatment
  Perceived intervention convenience will be benchmarked as an average score of ≥75 from a 0-100 scale.
Acceptability - Perceived Intervention Side Effects | Enrollment to end of 8-week treatment
  Perceived intervention side effects will be benchmarked as an average score of ≥75 from a 0-100 scale.
Acceptability - Appropriateness of Intervention Length and Frequency | Enrollment to end of 8-week treatment
  Appropriateness of intervention length and frequency will be benchmarked as an average score of ≥75 from a 0-100 scale.
Acceptability - Appropriateness of Daily Diary Length and Frequency | Enrollment to end of 8-week treatment
  Appropriateness of daily diary length and frequency will be benchmarked as an average score of ≥75 from a 0-100 scale.
Acceptability - Appropriateness of Other Study Measures | Enrollment to end of 8-week treatment
  Appropriateness of other study measures will be benchmarked as an average score of ≥75 from a 0-100 scale.

OTHER OUTCOMES:
Pain Severity | Enrollment to end of 3-month follow-up
  The Brief Pain Inventory (BPI) will be incorporated into daily diary assessment which will be completed by participants once per day for 7 consecutive days at four key time points: (1) baseline (prior to intervention exposure), (2) mid-treatment (at week 4), (3) immediate post-treatment, and (4) the 3-month follow-up. Pain severity will be determined by the mean of four BPI items (i.e., "average," "worst," "least" pain experienced in the past 24 hours, and pain experienced "right now"). All of these items are measured on a 0 to 10 Numerical Rating Scales (0 = "No pain", 10 = "Pain as bad as you can imagine").
Pain Interference | Enrollment to end of 3-month follow-up
  The Brief Pain Inventory (BPI) will be incorporated into daily diary assessment which will be completed by participants once per day for 7 consecutive days at four key time points: (1) baseline (prior to intervention exposure), (2) mid-treatment (at week 4), (3) immediate post-treatment, and (4) the 3-month follow-up. Pain interference will be assessed by computing the mean of seven items that evaluate the extent to which an individual's pain has interfered with their general activity, mood, walking ability, normal work, relationship with others, sleep, and enjoyment of life within the past 24 hours. All of these items are measured on a 0 to 10 Numerical Rating Scales (0 = "No pain", 10 = "Pain as bad as you can imagine").
Physical Functioning | Enrollment to end of 3-month follow-up
  The PROMIS Short Form v2.0 - Physical Function 8b will be incorporated into online, self-reported assessments delivered via REDCap which will be completed by participants at four key time points: (1) baseline (prior to intervention exposure), (2) mid-treatment (at week 4), (3) immediate post-treatment, and (4) the 3-month follow-up. Physical functioning will be assessed as the function of upper and lower extremities, central core regions, and the ability to complete daily activities on a 5-point Likert scale.
Depression | Enrollment to end of 3-month follow-up
  The PROMIS Short Form v1.0 - Depression 8a will be incorporated into online, self-reported assessments delivered via REDCap which will be completed by participants at four key time points: (1) baseline (prior to intervention exposure), (2) mid-treatment (at week 4), (3) immediate post-treatment, and (4) the 3-month follow-up. Depression will be assessed by computing the mean of eight items that evaluate the extent to which depression-related symptoms are present on a 5-point Likert scale.
Anxiety | Enrollment to end of 3-month follow-up
  The PROMIS Short Form v1.0 - Anxiety 8a will be incorporated into online, self-reported assessments delivered via REDCap which will be completed by participants at four key time points: (1) baseline (prior to intervention exposure), (2) mid-treatment (at week 4), (3) immediate post-treatment, and (4) the 3-month follow-up. Anxiety will be assessed by computing the mean of eight items that evaluate the extent to which anxiety-related symptoms are present on a 5-point Likert scale.
Opiod Use | Enrollment to end of 3-month follow-up
  Questions pertaining to opioid analgesic us will be incorporated into daily diary assessment which will be completed by participants once per day for 7 consecutive days at four key time points: (1) baseline (prior to intervention exposure), (2) mid-treatment (at week 4), (3) immediate post-treatment, and (4) the 3-month follow-up. Opioid use will be assessed with various questions asking opioid use-related questions, including the frequency and dose.
Patient Global Impression of Change | Enrollment to end of 3-month follow-up
  The Patient Global Impression of Change measure will be incorporated into online, self-reported assessments delivered via REDCap which will be completed by participants at four key time points: (1) baseline (prior to intervention exposure), (2) mid-treatment (at week 4), (3) immediate post-treatment, and (4) the 3-month follow-up. Belief of treatment efficacy will be assessed by computing the mean of seven items that evaluate the extent to which a participant believes their symptoms have improved on a 7-point Likert scale ranging from "very much improved," "much improved," "minimally improved," "no change," "minimally worse," "much worse," to "very much worse".
Mindfulness | Enrollment to end of 3-month follow-up
  The Mindful Attention Awareness Scale (MAAS) will be incorporated into online, self-reported assessments delivered via REDCap which will be completed by participants at four key time points: (1) baseline (prior to intervention exposure), (2) mid-treatment (at week 4), (3) immediate post-treatment, and (4) the 3-month follow-up. Mindfulness will be assessed by computing the mean of 15 items that evaluate the extent to which a participant is mindful throughout daily activities on a 6-point Likert scale ranging from "almost always," to "almost never".
Pain Catastrophizing | Enrollment to end of 3-month follow-up
  The Pain Catastrophizing Scale (PCS) will be incorporated into online, self-reported assessments delivered via REDCap which will be completed by participants at four key time points: (1) baseline (prior to intervention exposure), (2) mid-treatment (at week 4), (3) immediate post-treatment, and (4) the 3-month follow-up. Pain catastrophizing will be assessed by computing the mean of 13 items that evaluate the extent to which a participant engages in pain-related thoughts on a 5-point Likert scale ranging from "not at all," to "all the time".
Insomnia Symptoms | Enrollment to end of 3-month follow-up
  The Insomnia Severity Index (ISI) will be incorporated into online, self-reported assessments delivered via REDCap which will be completed by participants at four key time points: (1) baseline (prior to intervention exposure), (2) mid-treatment (at week 4), (3) immediate post-treatment, and (4) the 3-month follow-up. Insomnia will be assessed by computing the mean of seven items that evaluate the extent to which a participant experiences insomnia symptoms on a 5-point Likert scale ranging from "none/not at all," to "very/very much".
Conditioned Pain Modulation | Enrollment to end of 8-week treatment
  Conditioned pain modulation (CPM) will be assessed using Quantitative Sensory Testing and will be delivered at three key time points: (1) baseline (prior to intervention exposure), (2) mid-treatment (at week 4), and (3) immediate post-treatment. Endogenous pain inhibition is assessed by the CPM index. A CPM Index will be quantified as the average percent change in pressure pain threshold during cold pressor task relative to the baseline pressure pain threshold.
Adverse Events | Enrollment to end of 3-month follow-up
  Reports of adverse events will be monitored throughout the study period for all study participants.

CONTACTS AND LOCATIONS:
Overall Officials: Chung Jung Mun, PhD, Principal Investigator — Arizona State University
Locations (2):
- United States (2):
  - Arizona State University Downtown Phoenix Campus, Phoenix, Arizona
  - Arizona State University, Phoenix, Arizona

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Mun CJ, Contreras E, Xiao Y, Eckert R, Harting A, Damera S, Perez I, Pandey HK, Mardian AS, LoVecchio F, Colloca L, Dunn KE, Todd M, Fillingim RB, Davis MC. Combining mindfulness intervention and open-label placebo treatment for chronic pain: a protocol for a feasibility study. Pilot Feasibility Stud. 2025 Aug 20;11(1):111. doi: 10.1186/s40814-025-01692-8. PMID 40836262